CLINICAL TRIAL: NCT02901327
Title: Effects of Lumbar Stabilisation Exercise and Treadmill Walk on Multifidus Activation, Pain and Functional Disability in Individuals With Chronic Low Back Pain
Brief Title: Multifidus Activation, Pain and Functional Disability in Individuals With Chronic Low Back Pain
Acronym: CMLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayero University Kano, Nigeria (Other)
Responsible Party: Principal Investigator, BASHIR BELLO, Dr., Bayero University Kano, Nigeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BayeroUK
Record Dates: First submitted 2016-06-09; First posted 2016-09-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Low Back Pain
Keywords: Lumbar Stabilisation Exercise; Treadmill Walk; Multifidus Muscle Activation; Pain Intensity; Functional Disability
MeSH Terms: conditions — Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar Stabilisation Exercise (Experimental): 30 minute lumbar stabilization exercise, 3 times per week for 8 weeks.
  Interventions: Procedure: Lumbar Stabilisation Exercise
- Treadmill walk exercise (Active Comparator): Walking exercise on a treadmill for a maximum of 30 minutes with increasing speed and inclination. 3 times/week for 8 weeks.
  Interventions: Procedure: treadmill walk exercise

INTERVENTIONS:
Procedure: Lumbar Stabilisation Exercise — McGill protocol starting with:
  1. 'cat-camel' exercise exercise 10 repetitions with 7 seconds hold each
  2. 'curl-up' exercise 10 repetitions with 7 seconds hold each
  3. 'side-bridge' exercise 10 repetitions with 7 seconds hold each
  4. 'cat-camel' exercise 10 repetitions with 7 seconds hold each progression was based on subjects' tolerance and endurance.
  Other Names: Core Exercise
  Arms: Lumbar Stabilisation Exercise
Procedure: treadmill walk exercise — Bruce protocol
  This include:
  1. '5 minutes warm up' at zero degree inclination.
  2. '20 minutes active exercise with increasing speed and inclination'
  3. '5 minutes cool down'
  Other Names: Aerobic Exercise
  Arms: Treadmill walk exercise

SUMMARY:
Chronic Mechanical Low Back Pain (CMLBP) is a common disabling health problem among the general population. Multifidus muscle inhibition accompanying CMLBP plays a major role in perpetuating the pain and functional disability. Lumbar stabilisation and treadmill exercises are established treatments for CMLBP. However, it is not known which of the two techniques is more effective. This study was conducted to compare the effects of lumbar stabilisation and treadmill walk on multifidus activation, pain and functional disability in individuals with CMLBP.

DETAILED DESCRIPTION:
Fifty-three individuals (23 females and 30 males) with CMLBP participated in this single blind randomised clinical trial. Consecutive participants were recruited from the outpatient Physiotherapy clinic of the Aminu Kano Teaching Hospital, Kano, Nigeria and were randomly assigned to one of two exercise groups: Lumbar Stabilisation Group (LSG; n = 27) or Treadmill Walk Group (TWG; n = 26). However, 50 participants, (LSG: n = 25; and TWG: n = 25) completed the eight week study. Participants in the LSG had lumbar stabilisation exercises using McGill protocol while those in the TWG had walking exercise on a treadmill using the Bruce protocol. Treatment was applied three times weekly for eight weeks. Outcomes assessed at baseline and end of eighth week of study were: Pain Intensity (PI) using Visual Analogue scale, Functional Disability (FD) using Oswestry Disability Index Questionnaire; and Multifidus Muscle Activation (MMA) level using a surface electromyography machine. Data were analysed using descriptive statistics, paired and independent t-tests at α0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed with LBP of mechanical origin and have been present for 3 months or more.
2. Participants who have a score of at least 20% on Modified Oswestry Dis¬ability Index (ODI).
3. Participants who gave consent to participate in the study.
4. Participants who can comprehend instructions in English or Hausa
5. Participants who are not involved in any other form of exercise training during the course of the study.

Exclusion Criteria:

1. Patients with history of a prior surgery to the lumbosacral spine.
2. Patients with any neurological findings indicating radiculopathy.
3. Patients with very acute symptoms of LBP.
4. Patients with evidence of systemic disease, carcinoma or organ diseases.
5. Patients with obesity which due to reduce fatty infiltration that might affect electrical conductivity in the multifidus muscle.
6. Patients below 18 years of age.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Amplitude of Multifidus Muscle Activation | 8 weeks of intervention
  using the surface electromyography

SECONDARY OUTCOMES:
Functional Disability status | Baseline
  using the modified Oswestry disability index questionnaire
Functional Disability status | 8 weeks
  using the modified Oswestry disability index questionnaire
Pain Intensity | Baseline
  using the VAS
Pain Intensity | 8 weeks
  using the VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Kano State, Nigeria

IPD SHARING:
Plan to Share IPD: No